CLINICAL TRIAL: NCT02535845
Title: Developing a Self-persuasion Intervention Promoting Adolescent HPV Vaccination
Brief Title: Developing a Self-persuasion Intervention Promoting Adolescent HPV Vaccination: Feasibility Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Halted early due to poor accrual and lack of time to receive intervention procedures adjacent to a clinic visit post randomization.
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Southern Methodist University (Other); Parkland Health and Hospital System (Other)
Responsible Party: Principal Investigator, Jasmin A. Tiro, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01CA178414-04;STU 022013-016; 1R01CA178414 (NIH)
Record Dates: First submitted 2015-08-26; First posted 2015-08-31 (Estimated); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Human Papillomavirus Vaccines

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-persuasion group (Experimental): HPV information plus self-persuasion intervention in a tablet-based application (Project Voice)
  Interventions: Behavioral: Project Voice
- Information only group (Active Comparator): HPV information only in a tablet-based application (HPV Informational Video)
  Interventions: Behavioral: HPV Informational Video

INTERVENTIONS:
Behavioral: Project Voice — Project Voice tablet-based intervention plus informational video
  Arms: Self-persuasion group
Behavioral: HPV Informational Video — Informational video only
  Arms: Information only group

SUMMARY:
HPV vaccine coverage among adolescents in the US is suboptimal. This is particularly true among traditionally underserved adolescents. Few parent-targeted interventions have focused on the parental decision-making process. Self-persuasion, generating one's own arguments for engaging in a behavior, may be an effective means to influence parents' motivation to vaccinate their children. In a three-phase study, investigators are using quantitative and qualitative research methods to develop and refine a tablet-based self-persuasion intervention for parents who are undecided about the HPV vaccine. This clinical trial submission focuses on the third phase of the study (the second stage is also registered in clinical trials).

DETAILED DESCRIPTION:
Despite the fact that HPV vaccination is recommended for male and female adolescents, HPV vaccine coverage among adolescents age 13-17 is poor (60% for girls, 41.7% for boys). HPV-related cancers are a significant burden on the US healthcare system and could be prevented through adolescent vaccination. Rates of vaccination are suboptimal among underserved populations (uninsured, low-income, racial and ethnic minorities) often seen in safety-net clinics. Few interventions have been designed that target decision-making among parents of unvaccinated adolescents. Self-persuasion, generating of one's own arguments for a health behavior, may be an effective means of influencing HPV vaccination behaviors among undecided or ambivalent parents. Through three stages, investigators will identify and develop a self-persuasion intervention strategy to promote adolescent HPV vaccination in safety-net clinics. In Stage 3, reported here, investigators will conduct a two-arm pilot randomized control trial in the safety-net clinics to assess feasibility of testing the self-persuasion intervention condition against standard of care (control group). Parent-adolescent child dyads will be enrolled. Parents will be exposed to the intervention and the primary outcome (HPV vaccination) will be assessed on the adolescent child via the electronic health record. Investigators will also examine the impact of the intervention on parent-provider discussions about HPV vaccination.

ELIGIBILITY:
Inclusion Criteria for the Parent-Adolescent Dyad:

* Parents: Undecided about the HPV vaccine
* Adolescent child: 11-17 years old and has not begun the HPV vaccine series.

Exclusion Criteria:

* Parents: Having impairing hearing or speech
* Adolescents: pregnant at the time of the clinic visit
* Dyad: participated in Phase 1 and 2 of the study

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jasmin A Tiro, PhD, Principal Investigator — University of Texas Southwestern Medical Center; Austin S Baldwin, PhD, Principal Investigator — Southern Methodist University
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Tiro JA, Lee SC, Marks EG, Persaud D, Skinner CS, Street RL, Wiebe DJ, Farrell D, Bishop WP, Fuller S, Baldwin AS. Developing a Tablet-Based Self-Persuasion Intervention Promoting Adolescent HPV Vaccination: Protocol for a Three-Stage Mixed-Methods Study. JMIR Res Protoc. 2016 Jan 29;5(1):e19. doi: 10.2196/resprot.5092. PMID 26825137

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Parent-adolescent dyads were randomized to intervention arms. Parents were exposed to the intervention arm. Primary outcome measure (HPV vaccination) was assessed on the adolescent child via the electronic health record. The number started/completed represents the number of parent-adolescent dyads.
Groups:
- Self-persuasion Group - Parent: HPV information plus self-persuasion intervention in a tablet-based application (Project Voice)
  Project Voice: Project Voice tablet-based intervention plus informational video
- Self-persuasion Group - Adolescent: Adolescent's parent was exposed to HPV information plus self-persuasion intervention in a tablet-based application (Project Voice)
  Project Voice: Project Voice tablet-based intervention plus informational video
- Information Only Group - Parent; Information Group Only - Adolescent: HPV information only in a tablet-based application (HPV Informational Video)
  HPV Informational Video: Informational video only
Period: Overall Study
Arm/Group | Self-persuasion Group - Parent | Self-persuasion Group - Adolescent | Information Only Group - Parent | Information Group Only - Adolescent
Started | 7 | 7 | 4 | 4
Completed | 7 | 7 | 4 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Self-persuasion Group-Parent: HPV information plus self-persuasion intervention in a tablet-based application (Project Voice)
  Project Voice: Project Voice tablet-based intervention plus informational video
- Self-persuasion Group- Adolescent: Parent exposed to HPV information plus self-persuasion intervention in a tablet-based application (Project Voice)
  Project Voice: Project Voice tablet-based intervention plus informational video
- Information Only Group - Adolescent: Parent exposed to HPV information only in a tablet-based application (HPV Informational Video)
  HPV Informational Video: Informational video only
- Total: Total of all reporting groups
Arm/Group | Self-persuasion Group-Parent | Self-persuasion Group- Adolescent | Information Only Group - Parent | Information Only Group - Adolescent | Total
Number analyzed (Participants) | 7 | 7 | 4 | 4 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 7 | 0 | 4 | 11
  Between 18 and 65 years | 7 | 0 | 4 | 0 | 11
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 4 | 2 | 15
  Male | 0 | 5 | 0 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 1 | 1 | 10
  Not Hispanic or Latino | 3 | 3 | 3 | 3 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 3 | 3 | 12
  White | 4 | 4 | 1 | 1 | 10
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: HPV Vaccination Behavior Documented in Electronic Health Record, Initiation
Description: Number of parents who decided to start the HPV vaccine three dose series and got their child vaccinated within 30 days of the study appointment as evidenced by documentation in the child's electronic medical record.
Time Frame: 30 days
Population: Data were not collected due to early termination of the study
Groups:
- Self-persuasion Group - Adolescent: Parent exposed to HPV information plus self-persuasion intervention in a tablet-based application (Project Voice)
  Project Voice: Project Voice tablet-based intervention plus informational video
Arm/Group | Self-persuasion Group - Parent | Self-persuasion Group - Adolescent | Information Only Group - Parent | Information Only Group - Adolescent
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: HPV Vaccination Behavior Documented in Electronic Medical Record, Completion
Description: Number of doses received and the dates of those doses within 15 months of the study appointment as evidenced by documentation in the child's electronic medical record.
Time Frame: 15 months
Population: Data were not collected due to early termination of the study
Arm/Group | Self-persuasion Group | Information Only Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Active Parent Participation During Clinical Encounter
Description: Investigators will explore the factors associated with parent degree of participation in the discussion with the healthcare provider during the clinical encounter using Street coding scheme of 3 types of active communication.
Time Frame: 1 day
Population: Data were not collected due to early termination of the study
Arm/Group | Self-persuasion Group | Information Only Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Day of visit (1 day)
Description: Adverse event definitions are the same as clinicaltrials.gov definitions.
Groups:
- Self-persuasion Group - Parents; Self-persuasion Group - Adolescents: HPV information plus self-persuasion intervention in a tablet-based application (Project Voice)
  Project Voice: Project Voice tablet-based intervention plus informational video
- Information Only Group-Parents; Information Only Group - Adolescents: HPV information only in a tablet-based application (HPV Informational Video)
  HPV Informational Video: Informational video only
Arm/Group | Self-persuasion Group - Parents | Self-persuasion Group - Adolescents | Information Only Group-Parents | Information Only Group - Adolescents
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT02535845/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT02535845/ICF_001.pdf